CLINICAL TRIAL: NCT01871051
Title: Risk Factors For Postoperative Respiratory Complications After Anesthesia
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-4414
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project was aimed to identify the risk factors associated with the occurrence of respiratory complications in post anesthesia care unit. The primary outcome was the composite measure of occurrence of complications in PACU. The components were apnea or hypopnea, laryngospasm, bronchospasm and prolonged oxygen requirement.

DETAILED DESCRIPTION:
This is a retrospective project. Data will be used from Quality Improvement database for publication purpose. Data was collected from a prospectively collected database that was done as a Quality Improvement Project. The study sites included post anesthesia care units (PACU) of the main and ambulatory campuses of our hospital. The data was collected from surgical and radiology PACU's. Data was collected each quarter for 2 weeks in the surgical PACU, and for 1 month in Radiology PACU, from Sep 2007 through Mar 2012. Trained perioperative nurses and Certified Registered Nurse Anesthesiologist did data collection. This ensured a sample representative of at least 10% of patients anesthetized for surgical and radiological procedures. The independent variables (risk factors) collected included age, American Society of Anesthesiology (ASA) physical status, obesity, preexisting airway or lung disease, preexisting neuromuscular disease or hypotonia, morbid obesity, intraoperative bronchospasm and intraoperative laryngospasm. The primary outcome variables collected were Apnea or hypopnea, Laryngospasm, Bronchospasm, and prolonged Oxygen requirement. Apnea or hypopnea was defined by the need for bag mask ventilation, Laryngospasm by the requirement of a positive pressure ventilation of > 20 cmH2O or administration of succinylcholine, Bronchospasm by use of albuterol, and Oxygen requirement by continued oxygen administration to maintain SpO2>92% for 2 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1) All patients who receive an anesthetic in participating institutions who are under 18 years of age and where an anesthetic record is generated will be included in the overall statistics for each center -

Exclusion Criteria:

1) Patients older than 18 years of age.-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients who receive an anesthetic in participating institutions who are under 18 years of age and where an anesthetic record is generated will be included in the overall statistics for each center
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of complications in PACU | 4 years
  This project was aimed to identify the risk factors associated with the occurrence of respiratory complications in post anesthesia care unit. The primary outcome was the composite measure of occurrence of complications in PACU. The components were apnea or hypopnea, laryngospasm, bronchospasm and prolonged oxygen requirement.

SECONDARY OUTCOMES:
Improve the quality of care for children undergoing anesthesia | 4 years
  * To improve the quality of care for children undergoing anesthesia in the United States by identifying preventable causes of anesthesia and surgery-related adverse events.
  * To use root cause analysis to investigate significant adverse events.